CLINICAL TRIAL: NCT06065202
Title: Personalized Targeted Nutrition Via StructurEd Nutrition Delivery Pathway to Improve Recovery of Physical Function in Trauma
Brief Title: Personalized Nutrition to Improve Recovery in Trauma
Acronym: SeND Home
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112343
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Abdominal Trauma
Keywords: precision nutrition; critical care; trauma; parenteral nutrition; indirect calorimetry
MeSH Terms: conditions — Abdominal Injuries; Wounds and Injuries; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SeND Home Pathway (Experimental): Total parenteral nutrition (TPN) will begin within 72 hours of abdominal surgery. Calorie needs will be determined by indirect calorimetry. Nutritional shakes will begin when a liquid diet is started. These will be taken 3 times a day while in the hospital and for 4 weeks after discharge.
  Interventions: Dietary Supplement: Nutrition Supplement
- Standard Nutrition (No Intervention): Standard nutrition as determined by clinical providers.

INTERVENTIONS:
Dietary Supplement: Nutrition Supplement — Total parenteral nutrition (TPN) will be administered within 72 hours of abdominal surgery. Nutritional shakes will be started with a liquid diet and given 3 times a day. This will continue for 4 weeks after discharge.
  Other Names: CLINIMIX E 8/14 sulfite-free; CLINOLIPID 20%; Nutritional shakes
  Arms: SeND Home Pathway

SUMMARY:
The purpose of this study is to determine if a particular method of providing nutrition improves the outcomes of patients in the intensive care unit (ICU) who have undergone abdominal surgery following trauma and would require nutrition delivered via the bloodstream (called total parenteral nutrition or TPN). The nutrition method being tested is a structured nutrition delivery plan, called the SeND Home pathway, that involves TPN, oral nutrition supplements, and the use of a device (called an indirect calorimeter or IC) to measure calorie needs. Participants will be randomly assigned (like the flip of a coin) to the SeND Home program or standard of care nutrition. In the SeND Home program, participants will receive TPN, followed by oral nutrition supplements (shakes) for 4 weeks after discharge. The control group will follow standard of care nutrition delivery that begins during ICU stay and concludes at hospital discharge. Participants in both groups will undergo non-invasive tests that measure how much energy (calories) they are using, body composition, and muscle mass and complete walking and strength tests, and surveys about quality of life.

DETAILED DESCRIPTION:
Severe abdominal trauma can impact patients in a variety of ways. Current data shows that trauma patients can experience problems with physical function, muscle weakness, and poor quality of life after they are released from the hospital. There is a critical need to improve nutrition in trauma patients with severe abdominal injuries to optimize the recovery process. The purpose of this study is to evaluate if the use of a planned nutrition delivery plan with early intravenous (IV) nutrition will improve outcomes. Participants will be randomly assigned 1:1, like flipping a coin, to the SeND Home program or routine care.

Participants in the standard of care program will receive standard nutrition delivery as determined by clinical care providers. This may include TPN.

Participants in the SeND Home program will receive TPN within 72 hours of abdominal surgery. Indirect calorimetry will be used to determine nutrition needs.Once participants are able to have a liquid diet they will receive nutrition shakes up to 3 times a day while in the hospital and for 4 weeks after discharge.

Participants will undergo tests to measure muscle mass, have blood draws, complete walking and strength tests, and surveys about quality of life. These tests will be done at several times throughout hospitalization and participants will be asked to return for a 3 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* 15+ years old
* Penetrating abdominal trauma requiring emergent major abdominal surgery
* Admitted to the surgical ICU
* Not expected to receive oral nutrition for 72 hours or more

Exclusion Criteria:

* Patients who are unable to ambulate at baseline
* Expected withdrawal of life-sustaining treatment within 48 hours
* Prisoners
* Positive pregnancy test for women of child bearing potential.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in six-minute walk distance (6 MWD) | 3 months
  Change in 6MWD from baseline to day 14 or hospital discharge will be compared between the two study arms

SECONDARY OUTCOMES:
Change in physical function | baseline, day 14 or hospital discharge, 3 and 6 months post-hospital discharge
  This will be measured by comparing the changes in physical function tests (4 meter walk, sit-to-stand) between the two study arms.
Change in muscle strength | baseline, hospital discharge, 3 and 6 months post-hospital discharge
  This will be measured by comparing the changes in grip and quad strength tests between the two study arms.
Change in muscle mass | baseline, hospital discharge, 3 and 6 months post-hospital discharge
  This will be measured by comparing changes in bioelectrical impedance analysis (BIA) between the two study arms.
Change in Quality of Life (QoL) | baseline, 3 and 6 months post-hospital discharge
  This will be measured by comparing changes in the EuroQoL-5 Dimension and 43-item Trauma Specific Quality of Life measurement between the two study arms.
Change in cognition | baseline, 3 and 6 months post-hospital discharge
  This will be measured by looking at changes in mental health and cognition via questionnaires.
Infection | hospital discharge, 3 and 6 months post-hospital discharge
  This will be measured by looking at the number of infections reported.
Length of Hospital/ICU stay | hospital discharge
  This will be measured by recording the length of hospital stay noted in the medical record.
Mortality rate | 6 months post-hospital discharge
  This will be measured by survival after 6 months.
Change in muscle mitochondrial metabolism | admission, day 14, and hospital discharge
  This will be measured by doing urine and blood tests.
Change in key resilience and inflammation biomarkers | admission, day 14, and hospital discharge
  This will be measured utilizing the Duke Pepper Panel which serves as a comprehensive set of biological indicators typically incorporating: hormones, inflammatory markers and genomic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, MD, Principal Investigator — Duke
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No